CLINICAL TRIAL: NCT05298540
Title: Feasibility and Acceptability of Home-based Computerised Cognitive Training After Cardiac Surgery
Acronym: FACCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 309731
Record Dates: First submitted 2022-03-07; First posted 2022-03-28 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Cognitive intervention; Cardiac surgery; Feasibility; Acceptability
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based computerised cognitive training (Experimental): Participants will be asked to complete 40 sessions (20 minutes / day, 5 days / week) of cognitive training over the 8-week intervention period (this will be assessed using automated data reports of user activity generated in collaboration with BrainHQ). Training will commence one week postoperatively to avoid the effects of sedatives, postoperative pain, sleep deprivation, and patient fatigue, and to improve adherence
  Interventions: Behavioral: Home-based computerised cognitive training with BrainHQ

INTERVENTIONS:
Behavioral: Home-based computerised cognitive training with BrainHQ — Participants will be registered for individual accounts to an online CCT program created by BrainHQ (Posit Science, San Francisco), that can be administered using their own computer or tablet. BrainHQ has been associated with improvements in memory, attention, and processing speed. The program will be customised to target domains thought to be deficient in the postoperative period and will include training in memory, attention, and processing speed. Specifically, the following six games have been selected: hear, hear (auditory memory and attention), to-do list training (working memory), divided attention (attention), target tracker (attention), double decision (useful field of view and visual processing speed), and eye for detail (visual processing speed and visual working memory). The exercises are adaptive, adjusting the application difficulty to the participants performance.

SUMMARY:
The aims of this study are to (1) evaluate the feasibility and acceptability of a home-based computerised cognitive training programme in the postoperative cardiac surgical population, and (2) estimate measures of precision about the mean and variance of cognitive outcome to inform sample size calculations for a subsequent efficacy study.

DETAILED DESCRIPTION:
Heart surgery is a common procedure for coronary heart disease (blocked or narrowed coronary arteries) and valve problems (narrowing or hardening of the heart valves). It is known that after surgery some patients experience problems with their 'cognitive health' - this includes aspects like memory problems, concentration, and attention. These cognitive health problems can last for several months and can have a considerable impact on patients, and their family.

Cognitive training (which means exercising the brain) has been shown to improve cognitive health in a number of patient groups including healthy older adults, patients with heart failure, and patients with mild cognitive impairment. The aim of this study is to find out if home-based computerised cognitive training (CCT) improves cognitive health after heart surgery.

Investigators will recruit adult (≥ 18 years) patients undergoing first time elective cardiac surgery, who are willing to engage with an online training programme, and due to the nature of the intervention, potential participants must have access to a computer or tablet and access to the internet.

Before surgery, a brief cognitive assessment will be carried out. Participants will be asked to complete 20 minutes of cognitive training exercises, 5 days per week, starting one week after their operation. A member of the research team will contact the patient once a week to check progress, to provide support, and to help with any technical issues.

After the 8-week CCT (brain training exercises) programme, a follow-up video call will be arranged. During this follow-up participants will complete a second cognitive assessment and a questionnaire to see how acceptable and helpful they found the brain training exercises.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old undergoing first time elective cardiac surgery
* Willing to engage with an online cognitive training programme
* Access to a computer or table with access to the internet.

Exclusion Criteria:

* Unwilling or unable to give written informed consent
* significant psychiatric or medical comorbidities where that condition might impact on cognitive function and affect their ability to participate.
* Inability to understand written and / or verbal English
* Those with motor symptoms that would impede their ability to complete the programme
* Those unwilling or unable to engage in a video call

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  Number of participants included from eligible patients; satisfactory recruitment defined as enrolment of ≥ 50% of eligible patients.
Study retention | 6 months
  Satisfactory retention rate ≥ 75% of participants completing the 8-week training programme
Recruitment target | 6 months
  The time required to meet the target recruitment of 30 patients
Feasibility of testing procedures | 6 months
  % of participants where outcome testing was completed
Feasibility of data collection methods | 6 months
  % of participants with complete data sets
Adherence to the intervention: number of sessions | 6 months
  Compliance to measure the feasibility of the study; the number of sessions completed out of the 40 planned sessions during the 8-week intervention
Adherence to the intervention: total time | 6 months
  Compliance to measure the feasibility of the study; the total time completed out of the planned 800 minutes during the 8-week intervention
Acceptability, by participant report | measured after the 8 week intervention (ie 8-10 weeks)
  The theoretical framework of acceptability (TFA) questionnaire has been adapted to this study, in collaboration with one of the TFA development team, to evaluate participants' perceptions of the intervention. The questionnaire was designed to inductively evaluate the retrospective acceptability of the intervention. The seven-item questionnaire will provide a five-point Likert scale reporting method in relation to their agreement statements, where the minimum value is 5 and maximum value is 35, with a higher score indicating higher acceptability.

SECONDARY OUTCOMES:
to estimate measures of precision about the mean and variance of cognitive outcome to inform sample size calculations for a subsequent efficacy study. | 6 months
  Cognitive function will be measured using the Montreal Cognitive Assessment (MoCA). The MoCA is a brief, 30-question test of global cognition, designed to detect mild cognitive impairment with a high degree of sensitivity and specificity. The MoCA takes approximately 10 minutes to administer, and will be measured upon enrolment and after the 8-week intervention. A score of 26 (out of 30) or higher is considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Bowden, MSc, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There are no plans to share the data consistent with ethics approvals and consent.